CLINICAL TRIAL: NCT06999525
Title: Use of Virtual Reality Technologies in Management of Anxiety and Discomfort During Endoscopy Procedure
Acronym: CARVENDO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP231304; 2025-A00550-49 (Registry Identifier: IDRCB)
Record Dates: First submitted 2025-04-25; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Endoscopy
Keywords: Endoscopy; Virtual reality technologies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- With virtual reality technologies (Experimental): Patients with virtual reality technologies during endoscopy procedure
  Interventions: Device: Therapeutic virtual reality headset (CRVT)
- Without virtual reality technologies (No Intervention): Routine procedure of endoscopy

INTERVENTIONS:
Device: Therapeutic virtual reality headset (CRVT) — Contribution of the use of a Therapeutic Virtual Reality Headset in the management of anxiety and discomfort in digestive endoscopy
  Arms: With virtual reality technologies

SUMMARY:
Digestive endoscopies are performed either for diagnostic purposes (e.g. suspicion of cancer or monitoring of chronic diseases) or for therapeutic purposes (treatment of digestive haemorrhage, removal of polyps, etc.).

Some endoscopies are performed under local anaesthetic, which can cause considerable anxiety in anticipation of the procedure and considerable discomfort during the procedure. Other endoscopies are performed under general anaesthetic for more extensive procedures on outpatients or inpatients. Anxiety prior to anaesthesia is likely to increase the perception of pain, increase the need for anaesthetic products and thus increase the time to complete awakening.

Complementary techniques such as hypnotherapy can be used before the operation, with proven effectiveness. But these techniques require dedicated and specifically trained staff, as well as additional time.

Virtual reality technologies, and in particular virtual reality headsets, allow instant immersion in a relaxing world. Therapeutic virtual reality headsets (TRVH) have been shown to be effective in reducing pre-operative anxiety and pain perception.

Our hypothesis is that the use of a CRVT could reduce the consumption of anaesthetic products, reduce anxiety, improve overall satisfaction and reduce the length of outpatient hospitalisation during digestive endoscopy procedures.

DETAILED DESCRIPTION:
This is a single-centre randomised controlled trial. The aim is to compare total propofol consumption between patients who have benefited from CRVT immersion and control patients.

All consecutive eligible patients will be informed of the study and invited to participate, by the prescribing physicians, in consultation or during hospitalisation as part of their care. The presentation of the research will also include a demonstration of the use of the CRVT in the digestive endoscopy department.

Patients who agree to take part will be included on the day of the procedure and randomised immediately afterwards by the doctor performing the endoscopy, in a 1:1 ratio, using a secure web server.

Patients randomised to the experimental arm will receive CRVT pre-operatively. Pre-operative anxiety (STAI) will be measured on two occasions: on arrival in the endoscopy department (at reception) and before the endoscopic procedure (in the endoscopy room).

Sedation will be provided by IV propofol only, by AIVOC. The depth of sedation will be monitored by measuring the bispectral index (BIS), with the aim of achieving a score of ≤ 75. Maintenance of sedation in the target zone will be achieved by adjusting the target concentration of AIVOC, with a BIS target of between 65 and 75. The time between the end of the procedure and actual awakening will be recorded in the endoscopy room.

Patient satisfaction (quantitative scale from 0 to 100) will be assessed in the outpatient department (during the pre-discharge visit). The time elapsed between the end of the procedure and discharge from the outpatient department will be recorded at the time of discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years (adult patients)
* Affiliated with a French social security system
* No legal protection measures (e.g., guardianship, curatorship)
* Scheduled for outpatient digestive endoscopy (upper or lower) under general anesthesia, level 1 (excluding biliary or interventional procedures)
* Medical indication for the endoscopic procedure established by a clinician

Exclusion Criteria:

* History of epilepsy
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
total propofol consumption | at day 1
  To compare total propofol consumption between patients who received CRVT immersion and control patients.

SECONDARY OUTCOMES:
Time of awakening | at day 1
  To compare the time to awakening after the end of the procedure between patients who received CRVT immersion and control patients.
patient satisfaction | at day 1
  To compare patient satisfaction with CRVT immersion with that of control patients.
  Questionnaire: Visual Analog Scale Patient satisfaction assessed using a 0-100 Visual Analog Scale (VAS) Patient satisfaction will be assessed using a visual analog scale ranging from 0 to 100, where higher scores indicate greater satisfaction (better outcome).
  This scale will evaluate the patient's experience regarding:
  * Pain
  * Nausea
  * Anxiety
  * Overall satisfaction The questionnaire will be administered in the outpatient unit prior to discharge
post-endoscopy anxiety assessement | at baseline and at day 1
  To compare pre- and post-endoscopy anxiety in CRVT-immersion patients with that in control patients.
  Outcome Measure Description:
  Anxiety will be evaluated using the State-Trait Anxiety Inventory - State subscale (STAI-YA), a validated self-report questionnaire composed of 20 items rated on a 4-point Likert scale.
  * Score range: 20 (low anxiety) to 80 (high anxiety)
  * Interpretation: Higher scores indicate greater anxiety (worse outcome)
  The questionnaire will be administered twice:
  * Timepoint 1 - Upon arrival in the endoscopy unit (baseline)
  * Timepoint 2 - Immediately after the endoscopic procedure (Day 1) The difference in STAI-YA scores before and after the procedure will be compared between patients in the CRVT group and those in the control group
Duration of hospitalization | at day 1
  To compare the duration of outpatient hospitalisation between the end of the procedure and discharge of patients who had undergone CRVT immersion with that of control patients

CONTACTS AND LOCATIONS:
Overall Officials: Thomas BAZIN, MD, PhD, Principal Investigator — CHU Ambroise Paré, APHP, France

IPD SHARING:
Plan to Share IPD: Undecided